CLINICAL TRIAL: NCT00490061
Title: A Multi-Institutional Phase II Study of Radiation and GW572016 (Lapatinib) for Patients With Stage III-IV Head and Neck Cancer Who Cannot Tolerate Concurrent Chemoradiotherapy.
Brief Title: Lapatinib and Radiation for Stage III-IV Head and Neck Cancer Patients Who Cannot Tolerate Concurrent Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual.
Sponsor: Quynh-Thu Le (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Quynh-Thu Le, Professor Radiation Oncology, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENT0020; 97864 (Other: Stanford University Alternate IRB Approval Number); LAP #109855 (Other: GlaxoSmithKline); 8857 (Other: Stanford IRB)
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Head and Neck Cancer; Carcinoma, Squamous Cell; Head and Neck Cancers
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — Lapatinib; halofantrine; Radiotherapy; Radiation; Dynamic Contrast Enhanced Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiotherapy and Lapatinib with DCE-MRI (Experimental): DCE-MRI will precede radiotherpy before and after Lapatinib loading. 1500mg/d once daily oral Lapatinib will be administration for seven days prior to and throughout radiotherapy. Radiotherapy will be delivered as Intensity Modulated Radio Therapy (IMRT) using a G.E. Healthcare 1.5T MR, systems revision 12.0 M5 for a total dose of 70Gy delivered in 2-2.12 Gy/ fraction over the course of 6.5-7 weeks.
  Interventions: Drug: Lapatinib; Procedure: Radiotherapy (radiation); Device: G.E. Healthcare 1.5T MR, systems revision 12.0 M5; Device: DCE-MRI

INTERVENTIONS:
Drug: Lapatinib — 1500 mg po daily orally
  Other Names: Tykerb/Tyverb; GlaxoSmithKline
Procedure: Radiotherapy (radiation) — Standard of Care
  Other Names: IMRT - Intensity Modulated Radiotherapy
Device: G.E. Healthcare 1.5T MR, systems revision 12.0 M5 — Standard of Care, used to deliver IMRT
  Other Names: G.E. Healthcare MRI Device and Software
Device: DCE-MRI — A subset of patients received imaging before and after Lapatinib loading, prior to starting radiotherapy.
  Other Names: Dynamic contrast-enhanced magnetic resonance imaging

SUMMARY:
We propose to combine lapatinib with RT alone in patients with locally advanced head and neck cancer who cannot tolerate chemotherapy. The main objective of the study is to determine the efficacy of combining concurrent radiation and lapatinib in terms of time-to-progression (TTP) in this group of patients. In addition, we will determine the 2-year locoregional control rate (LRC), progression-free survival (PFS) and overall survival (OS) in these patients. We will also evaluate the profile and frequency of late toxicity, specifically mucosal and dermatologic toxicity, of the combination of lapatinib and RT in patients with locally advanced head and neck squamous cell carcinoma (HNSCC).

DETAILED DESCRIPTION:
There is substantial data to suggest that EGFR and Her-2/neu expressions are important predictors for prognosis in HNSCC. EGFR blockade with a monoclonal antibody in conjunction with radiotherapy has been shown to improve survival over radiotherapy alone in patients with locally advanced HNSCC. Dual inhibition of EGFR and ErbB2 tyrosine kinases results in greater inhibitory effect of the downstream signaling pathways in cancer cells than inhibition of either receptor alone. Phase I studies in HNSCC suggested that the drug is well tolerated when delivered either alone or concurrently with cisplatin based chemoradiotherapy in HNSCC.

We propose to combine lapatinib with RT alone in patients with locally advanced HNSCC who cannot tolerate chemotherapy. The main objective of the study is to determine the efficacy of combining concurrent radiation and lapatinib in terms of time-to-progression (TTP) in this group of patients. In addition, we will determine the 2-year locoregional control rate (LRC), progression-free survival (PFS) and overall survival (OS) in these patients. We will also evaluate the profile and frequency of late toxicity, specifically mucosal and dermatologic toxicity, of the combination of lapatinib and RT in patients with locally advanced HNSCC.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed stage III-IV HNSCC, pathologically confirmed (HNSCC from unknown primary sites are allowed)
* No evidence of distant metastasis
* No prior radiation therapy to the head and neck sites.
* Able to sign a study-specific informed consent form.
* Women of childbearing potential and men with partners capable of producing offspring must be willing to practice acceptable methods of birth control to prevent pregnancy.
* Left ventricular ejection fraction (LVEF) within the institutional normal range as measured by ECHO (If ECHO cannot be performed or if the Investigator feels that it is not conclusive to evaluate LVEF, then a MUGA scan should be performed).
* Having one of the following parameters that would preclude the use of concurrent CRT:

  * ECOG PS > 2.
  * Creatinine > 1.3 or calculate or measure creatinine clearance < 60 ml/min.
  * AST or ALT > 1.5 times normal limit but < 3 times normal limit
  * Total bilirubin > 1.5 mg/dL but < 3mg/dL
  * History of hearing loss that would preclude cisplatin chemotherapy. These would include the existing need of a hearing aid or a >= 25 decibel shift over 2 contiguous frequencies on a pretreatment hearing test.
  * Pre-existing peripheral neuropathy that would preclude cisplatin chemotherapy
  * Refuse or cannot tolerate chemotherapy
* Age 18 years or older

Exclusion Criteria:

* Known hypersensitivity to lapatinib or any of the excipients of this product (quinazolines).
* Uncontrolled angina, arrhythmia or congestive heart failure at the time of HNSCC diagnosis and treatment.
* History of myocardial infarction < 6 months from study entry.
* Treatment with a non-approved or investigational drug within 30 days before Day 1 of study treatment.
* Prior treatment with EGFR or Her2/Neu directed therapies.
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with Lapatinib.
* Absolute neutrophil count < 1500/uL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-07; Primary Completion 2013-01 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Quynh-Thu Le, Principal Investigator — Stanford University
Locations (5):
- United States (5):
  - Stanford University School of Medicine, Stanford, California
  - University of Florida Shands Cancer Center, Gainsville, Florida
  - Beth Israel, New York, New York
  - Duke University, Durham, North Carolina
  - University of Wisconsin Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place in a radiation oncology clinic, in a private room. The recruitment period spanned from 7/26/2007-11/18/2011.
Pre-assignment Details: # of subjects were screened.
Groups:
- Radiotherapy (Radiation) and Lapatinib: Lapatinib, 1500mg once daily, was administered for 7 days prior to, and for the duration of Intensity Modulated Radio Therapy (IMRT), delivered by G.E. Healthcare 1.5T MR, systems revision 12.0 M5 for a total dose of 70Gy delivered in 2-2.12 Gy/ fraction over the course of 6.5-7 weeks.
Period: Overall Study
Arm/Group | Radiotherapy (Radiation) and Lapatinib
Started | 17
Completed | 16
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Radiotherapy (Radiation) and Lapatinib: 1500mg/d once daily oral lapatinib administration plus Intensity Modulated Radio Therapy (IMRT) delivered by G.E. Healthcare 1.5T MR, systems revision 12.0 M5 for a total dose of 70Gy delivered in 2-2.12 Gy/ fraction over the course of 6.5-7 weeks.
  Lapatinib: 1500 mg po daily orally
  Radiotherapy (radiation): Standard of Care
  G.E. Healthcare 1.5T MR, systems revision 12.0 M5: Standard of Care, used to deliver IMRT
  PET/CT: A subset of patients received imaging before and after treatment.
Arm/Group | Radiotherapy (Radiation) and Lapatinib
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 13
Gender [Count of Participants; unit: Participants]
  Female | 5
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: To determine the efficacy of combining lapatinib and radiotherapy in terms of Progression-free survival (PFS) in patients with locally advanced HNSCC who cannot tolerate concurrent chemoradiotherapy.
  Progression-free survival is defined is the time from starting treatment to the time of first documented tumor progression or death due to any cause, which ever occurs first.
  Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST V1.0) as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 2 year PFS: PFS at 2 yrs after study enrollment
Population: All enrolled participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiotherapy (Radiation) and Lapatinib
Number analyzed (Participants) | 16
percentage of participants | 56.2 [47 to 65]

2. Secondary Outcome: Overall Survival.
Description: Overall survival is the time from starting treatment until death due to any cause. For subjects who do not die, time to death will be censored at the time of last contact.
Time Frame: Two years survival rate after study enrollment
Population: All enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Radiotherapy (Radiation) and Lapatinib
Number analyzed (Participants) | 16
percentage of participants | 62.5

ADVERSE EVENTS:
Time Frame: 2 years
Description: acute and late AE assessed at follow up appointments
Arm/Group | Radiotherapy (Radiation) and Lapatinib
Serious Adverse Events (participants affected / at risk) | 6/16
Other Adverse Events (participants affected / at risk) | 8/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiotherapy (Radiation) and Lapatinib (N=16)
Edema, larynx (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1 (1) — Bilateral pulmonary emboli
Hemolysis (Blood and lymphatic system disorders) | 1 (1) — Drug (baraclude) induced hemolytic anemia
ALT Increased (Investigations) | 1 (1) — Alanine aminotransferase increased
Lymphopenia (Immune system disorders) | 1 (1) — Lymphocyte count decreased.
Hyponatermia (Metabolism and nutrition disorders) | 1 (1) — Low concentration of sodium in the blood.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiotherapy (Radiation) and Lapatinib (N=16)
Elevated ALT (Investigations) | 2 (2) — Elevated alanine aminotransferase
Elevated AST (Investigations) | 3 (3) — Elevated aspartate aminotansferase
Elevated ALK (Investigations) | 2 (2) — Elevated Alkaline phosphatase
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — pneumonia
Dehydration (Metabolism and nutrition disorders) | 1 (1) — excessive loss of water
diarrhea (Gastrointestinal disorders) | 1 (1) — frequent and watery bowel movements
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) — Low concentrations of sodium in the blood

LIMITATIONS AND CAVEATS:
Due to low accrual, this study was terminated prior to reaching 60 subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No